CLINICAL TRIAL: NCT05280808
Title: Device Clinical Trial of the Efficacy of Using Novel Remote Self-fitting Software Compared With Standard Remote Fitting Software in the Customisation of Hearing-aid Settings for Adults With Hearing Loss
Brief Title: Evaluation of Software for Self-Fitting of Hearing Aids by People With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Sonova Audiological Care Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-385
Record Dates: First submitted 2022-02-23; First posted 2022-03-15 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental phone app (Experimental): Experimental phone app for self-fitting of hearing aids
  Interventions: Device: Experimental phone app used for self-fitting of hearing aids

INTERVENTIONS:
Device: Experimental phone app used for self-fitting of hearing aids — This software allows participants to set up hearing aids as appropriate for their hearing loss

SUMMARY:
The purpose of the study is to evaluate the efficacy of a prototype app for the self-fitting of hearing aids.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, clients giving written informed consent will be enrolled as participants. Each participant will use the app to self-fit and fine-tune the study aids over 30 days. Outcome measures include speech perception tests, questionnaires and the need for support with using the app. Own-aid performance is the reference, while unaided performance is the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Online client
* Daily aid use
* Bilateral aid use
* Uses P70-R or P90-R aids (same model both ears)
* Does not use earmolds
* Uses same soft tip on both aids
* Owns iPhone7/iOS12 or later
* Willing to install prototype app on own phone and use it in study
* Willing to participate in study for 30 days

Exclusion Criteria:

* Dexterity or cognitive issues that would be problematic for using the app in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Change in speech perception after 30 days | Day 1 and Day 30
  The online Speech Perception Test developed by Blamey Saunders Hearing will be used to assess the effect of the intervention on speech perception.
Change in self-rated hearing ability after 30 days | Day 1 and Day 30
  An expanded version of the Client Oriented Scale of Improvement questionnaire will be used to assess the effect of the intervention on self-rated hearing ability in different listening situations.
Softest sounds that can be heard | Day 1
  The intervention will be used to measure the softest sounds that can be heard at different tone frequencies.

SECONDARY OUTCOMES:
Change in preferences for fitted settings and fitting method over 30 days | Day 1, Day 10, Day 20 and Day 30.
  A custom questionnaire will be used to assess preferences for the fitted settings and fitting method of the intervention as these preferences evolve over time.
Change in experimental self-fitting phone app use over 30 days | Days 1-30
  The use of the experimental self-fitting phone app will be automatically logged every day to assess changes in how the app is used over time.

CONTACTS AND LOCATIONS:
Overall Officials: Justin A Zakis, PhD, Principal Investigator — Sonova Audiological Care Australia
Locations (1):
- Melbourne Support Office and Clinic/Teleaudiology, Carlton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No